CLINICAL TRIAL: NCT05576441
Title: Comparative Evaluation of Efficacy of Volume Stable Collagen Matrix in Interdental Papilla Reconstruction as Compared to Connective Tissue Graft in Maxillary Esthetic Region: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Volume Stable Collagen Matrix in Interdental Papilla Reconstruction in Maxillary Esthetic Region
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Geetanjali Sharma
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Gingival Recession Localized Moderate
Keywords: Interdental papilla reconstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group: VCMX (Experimental): Volume stable collagen matrix will be placed at recipient site and suturing will be done with a 5-0 vicryl suture.
  Interventions: Procedure: volume stable collagen matrix
- Control group:SCTG (Experimental): SCTG will be harvested from donor site as per the requirement and will be placed at the recipient and suturing will be done with 5-0 vicryl suture.
  Interventions: Procedure: subepithelial connective tissue graft

INTERVENTIONS:
Procedure: volume stable collagen matrix — Volume stable collagen matrix will be placed at recipient site and suturing will be done with a 5-0 vicryl suture.
  Arms: test group: VCMX
Procedure: subepithelial connective tissue graft — SCTG will be harvested from donor site as per the requirement and will be placed at the recipient and suturing will be done with 5-0 vicryl suture.
  Arms: Control group:SCTG

SUMMARY:
: Interdental papilla deficiency leads to food impaction, problems with phonetics and an unaesthetic appearance. Reconstruction of the deficient papilla is therefore, important. The purpose of study is to compare the VCMX and SCTG in papillae reconstruction. The null hypothesis is that there is no significant difference in clinical outcome for interdental papilla regeneration by volume stable collagen matrix and subepithelial connective tissue graft.

DETAILED DESCRIPTION:
The loss of interdental papillae can lead to formation of "black triangle/black holes" which may cause cosmetic, phonetics and functional problem(lateral food impaction).It may be due to plaque associated lesions, traumatic oral hygiene procedure, diverging tooth roots following orthodontic treatment, spacing between the teeth, abnormal tooth crown or contour of restoration.Surgical technique includes the pedicle graft procedure,envelop type flap using subepithelial connective tissue grafting(SCTG) or Platelet rich fibrin(PRF) at recipient site. A new volume stable cross linked collagen matrix (VCMX) is one such substitute for soft tissue regeneration.VCMX (fibrogide) is porcine, having only one porous layer which is made up of collagen having crosslinking to provide good volume stability and some elasticity at the same time. Porous layer promote angiogenesis, ingrowth of fibroblast, matrix biosynthesis and tissue integration. Main advantage is ability to maintain good volume stability. Apart from this less pain, less surgical chair time, faster wound healing as compared to connective tissue graft. VCMX shows promising results in term of volume gain, without any adverse reaction in various preclinical and clinical studies of soft tissue augmentation at implant sites.It also shows similar volume gain when augmenting implant sites with SCTG or VCMX. The purpose of study is to compare the VCMX and SCTG in papillae reconstruction. The null hypothesis is that there is no significant difference in clinical outcome for interdental papilla regeneration by volume stable collagen matrix and subepithelial connective tissue graft.

MATERIAL AND METHODS:

The present Prospective, analytical,Randomized Controlled clinical trial will be conducted in the Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences,Rohtak. In order to guarantee balance in patients allocated to either group ,block randomization will be used .Allocation concealment will be performed by a study monitor, preparing the assignment in opaque, sealed envelopes. Single blinding will be adopted where investigator analysing the result will be unaware to which group the patient belongs. Patient will be educated about the papillary recession and its implications. Scaling and root planing will be performed if needed. Thirty six Patients enrolled in the study will be randomly divided into two groups: TEST GROUP (n= 18) in which volume stable collagen matrix will be placed at the recipient site created by Han & Takei procedure in the deficient interdental papilla and CONTROL GROUP (n=18) in which subepithelial connective tissue graft will be harvested from donor site and placed at the recipient site created by Han & Takei procedure in the deficient interdental papilla. Patients will be re-evaluated for papillary fill after 1 month,3 months, 6 months respectively. Primary outcome measures includes Gain in papillary height in terms of distance measured from tip of papilla to an imaginary line connecting most apical point of gingival zenith of adjacent teeth. secondary outcomes include Full mouth indices Gingival Index (GI),Plaque Index (PI) Site specific Indices Gingival Index(GI), Plaque Index(PI), Papillary bleeding index ,Pocket Probing Depth (PPD), Clinical attachment loss(CAL), Width of keratinized gingiva(WKG), Distance from contact point to tip of papilla(CP-TP), Healing Index(HI)

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age range of 18-55 years who are systemically healthy.
* Patients with class II papillary recession according to Norland and Tarnow's classification and radiographically,the distance between contact point(CP) to alveolar crest ≤ 6mm.
* Patients who have completed etiological periodontal therapy(full mouth scaling and root planning)with Plaque index(Silness and Loe)<1,gingival index(Loe and silness)<1 and showing adequate compliance and willing to participate in the study.
* Patient complains of food lodgement or esthetic consideration for open gingival embrasure

Exclusion Criteria:

* Patients with the history of uncontrolled hypertension, diabetes,hyperthyroidism and on medications that influence the outcome of periodontal therapy.
* Presence of open contacts in the maxillary anterior region.
* Presence of crowding in the maxillary anterior region.
* Pregnant and lactating women.
* Patients with active periodontal disease
* Smokers,tobacco users

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Gain in papillary height | 6 months
  distance measured from tip of papilla to an imaginary line connecting most apical point of gingival zenith of adjacent teeth will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Sharma, BDS, Principal Investigator — Post graduate institute of dental sciences,Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India